CLINICAL TRIAL: NCT04916288
Title: Position of Puncture Point of the Introducer Needle During Internal Jugular Venous Catheterization With Ultrasound Guidance
Brief Title: Needle Puncture Point During Central Venous Catheterization With Ultrasound Guidance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Associate professor, Seoul National University Hospital
Other Study IDs: 10-2020-213
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Central Venous Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: central venous cathterization — central venous catheterization through the right internal jugular vein

SUMMARY:
In this observational study, we will measure the shortest distance from the cricoid cartilage level to the puncture site of the introducer needle when anesthesiologists perform central venous catheterization.

DETAILED DESCRIPTION:
After anesthesia induction and tracheal intubation, we will prepare central venous catheterization for patients requiring it. After anesthesiologists who are blinded to this study perform central venous catheterization, an investigator measured the shortest distance from the crease line of the cricoid cartilage to the puncture site of the introducer needle.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery under general anesthesia
* requirement of central venous catheterization

Exclusion Criteria:

* disagreement for participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years old) scheduled to elective surgery requiring central venous catheterization under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-08-16 (Estimated); Primary Completion 2022-07-16 (Estimated); Study Completion 2022-08-16 (Estimated)

PRIMARY OUTCOMES:
puncture site | intraoperative
  distance from the crease line of the cricoid cartilage to the puncture site of the introducer needle

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, MD.PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
If there would be a proper reason, I will share the data to other researchers.